CLINICAL TRIAL: NCT01623466
Title: A Randomized, Open-Label, Parallel Group Study To Evaluate Pharmacokinetic Profile, Wearability And Safety of Two Progestin-Only Patches Containing Different Doses Of Levonorgestrel (LNG)
Brief Title: Study to Evaluate Pharmacokinetics Profile, Wearability, and Safety of 2 Progestin-Only Patches
Acronym: ATI-CL21
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Agile Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATI-CL21
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Healthy
Keywords: PK and Safety
MeSH Terms: interventions — Levonorgestrel; Transdermal Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AG890-6.5 (Experimental): Evaluate levonorgestrel delivery in AG890-6.5
  Interventions: Drug: levonorgestrel
- AG890-12.5 (Experimental): Evaluate levonorgestrel delivery in AG890-12.5
  Interventions: Drug: levonorgestrel

INTERVENTIONS:
Drug: levonorgestrel — transdermal contraceptive delivery system
  Other Names: patch, transdermal contraceptive delivery system

SUMMARY:
Pharmacokinetics, safety and wearability in two size patches of AG890 over eight weeks will be evaluated.

DETAILED DESCRIPTION:
To evaluate pharmacokinetic (PK) profile, patch wearability (adhesion and skin irritation), and safety of AG890-6.5 and AG890-12.5 TCDS.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) greater than or equal to 18.
* Willing to use a non-hormonal method of contraception if of childbearing potential, or have already undergone previous bilateral tubal ligation or hysterectomy
* Willing to refrain from excessive use of alcohol from 48 hours prior to patch application through completion of the study.

Exclusion Criteria:

* Known or suspected pregnancy
* Lactating women
* Status post-partum or post-abortion within a period of 2 months prior to the start of study medication
* A cervical cytology smear of Papanicolaou (Pap) class III or greater or a Bethesda System report of low grade squamous intraepithelial lesions (SIL) or greater
* Smoking
* Hypertension (blood pressure >140 mm Hg systolic and/or >90 mm Hg diastolic)
* Valvular heart disease with complications
* ECG (in women with BMI ≥35 kg/m2) with clinically significant findings
* Diabetes Mellitus
* History of headaches with focal neurological symptoms
* Uncontrolled thyroid disorder
* Sickle cell anemia
* Current or history of clinically significant depression in the last year
* Known disturbance of lipid metabolism
* Acute or chronic hepatocellular disease with abnormal liver function
* Hepatic adenoma or carcinoma
* Cholestatic jaundice of pregnancy or jaundice with prior hormonal contraceptive use
* Plans for major surgery
* History of or existing venous and arterial thrombotic and thromboembolic disorder, vascular disease, cerebral vascular, or coronary artery disease
* Undiagnosed abnormal genital bleeding
* Known or suspected breast carcinoma, endometrial carcinoma, or estrogen-dependent neoplasia
* History or presence of dermal hypersensitivity in response to topical applications (bandages, surgical tape, etc.)
* Use of an injectable hormonal contraceptive within the past 10 months prior to the screening visit
* Use of a contraceptive implant or hormone-medicated intrauterine device (IUD) within 1 month prior to the screening visit
* Use of oral contraceptives or other sex steroid hormones within 2 months prior to the screening visit
* Chronic use of any medication that might interfere with the efficacy of hormone contraceptives (including barbiturates, bosentan, carbamazepine, felbamate, griseofulvin, oxcarbazepine, phenytoin, rifampin, St. John's Wort, topiramate, and HIV protease inhibitors), OR use of these medications within the past 3 months prior to screening visit
* A recent history (within prior 2 years ) of drug or alcohol abuse

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Garner, MD, PHD, Study Director — Agile Therapeutics

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AG890-6.5 | AG890-12.5
Started | 18 | 18
Completed | 17 | 18
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | AG890-6.5 | AG890-12.5 | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.83 (8.473) | 34.94 (6.673) | 32.39 (7.951)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Levonorgestrel Pharmacokinetic Profile
Description: The percentage of subjects with a minimal LNG level below pre-specified threshold of 175 pg/mL during the study.
Time Frame: 8 weeks
Population: Primary PK population
Measure: Number; unit: % of subjects below 175 pg/mL
Arm/Group | AG890-6.5 | AG890-12.5
Number analyzed (Participants) | 17 | 18
% of subjects below 175 pg/mL | 100 | 83.3

2. Primary Outcome: Evaluation of Patch Adhesion
Description: Evaluation of worst patch adhesion score for each subject using a 5-point adhesion scale:
  0: ≥90% adhered (no lift)
  1. ≥75% adhered but <90% (some edges showing lift)
  2. ≥50% adhered but <75% (half of system lifts off)
  3. <50% (< half of system lifts off, but undetached)
  4. patch completely detached
Time Frame: 8 weeks
Population: Safety population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AG890-6.5 | AG890-12.5
Number analyzed (Participants) | 17 | 18
Score on a scale | 0.41 (1.004) | 0.78 (1.517)

3. Primary Outcome: Evaluation of Irritation at Patch Application Site
Description: Self-reported worst skin irritation score at patch application site for each subject using a 4-point irritation scale:
  0: None
  1. Mild
  2. Moderate
  3. Severe
Time Frame: 8 weeks
Population: Safety population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AG890-6.5 | AG890-12.5
Number analyzed (Participants) | 18 | 18
Score on a scale | 0.11 (0.471) | 0.06 (0.236)

4. Primary Outcome: Evaluation of Itching at Patch Application Site
Description: Self-reported worst skin itching at patch application site by subject using a 4-point scale:
  0. None
  1. Mild
  2. Moderate
  3. Severe
Time Frame: 8 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | AG890-6.5 | AG890-12.5
Number analyzed (Participants) | 18 | 18
Score | 0.33 (0.594) | 0.39 (0.502)

5. Primary Outcome: Cycle Control
Description: Measurement of unscheduled bleeding/spotting days.
Time Frame: 8 weeks
Population: Completed subjects
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AG890-6.5 | AG890-12.5
Number analyzed (Participants) | 17 | 18
days | 8.4 (4.81) | 8.3 (4.23)

ADVERSE EVENTS:
Arm/Group | AG890-6.5 | AG890-12.5
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 11/18 | 9/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AG890-6.5 (N=18) | AG890-12.5 (N=18)
Gastrointestinal Disorders (Gastrointestinal disorders) | 1 (1) | 1 (2)
Immune system disorders (Immune system disorders) | 1 (1) | 0 (0)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Nervous system disorders (Nervous system disorders) | 9 (9) | 5 (5)
Psychiatric disorders (Psychiatric disorders) | 1 (1) | 2 (2)
Reproductive system ad breast disorders (Reproductive system and breast disorders) | 3 (3) | 5 (5)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications must be reviewed and approved by sponsor